CLINICAL TRIAL: NCT05563662
Title: SURgical Registry of Infective ENDocarditis in EuRope - SURRENDER
Brief Title: SURgical Registry of ENDocarditis EuRope
Acronym: SURRENDER
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Matthias Thielmann, Prof. Dr. med., University Hospital, Essen
Other Study IDs: WDHZ-TC-SURRENDER
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Infective Endocarditis; Cardiac Surgery; Outcomes
Keywords: Infective Endocarditis; Registry; European; Surgery; Prognosis
MeSH Terms: conditions — Endocarditis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgery — Patients with infective endocarditis undergoing open heart surgery

SUMMARY:
This is a prospective, multicentric, european registry of patients with infective endocarditis undergoing cardiac surgery. Patient demographics, clinical data and laboratory values will be collected, as well as treatment outcomes at day 30, day 90 and 1-5 years after the intervention.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is now a relatively rare but worldwide disease (3-10 IE/100000 population/year) with increasing incidence especially in the Western world. IE is still associated with high morbidity and mortality, prolonged hospital stay, high risk of reinfection, significantly worsened prognosis for patients, substantially reduced quality of life, and in any case represents a major financial burden for the respective healthcare systems [1-11].

Patients who need to undergo cardiac surgery due to infective endocarditis (IE) are heterogeneous and present with a persistently high perioperative morbidity and mortality rate. Despite optimal and individualized perioperative management strategies, perioperative complications such as heart failure, systemic inflammatory response, vasoplegia, and sepsis is still the main reason for adverse outcomes following cardiac surgery.

The present European, multicenter IE registry (Surgical RegistRy of infective ENDocarditis in EuRope - SURRENDER) was initiated and established to record and appropriately analyze current surgical treatment options and perioperative adjunctive treatment strategies, as well as short- and long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infective endocarditis (according to DUKE criteria) undergoing cardiac surgery
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Missing declaration of consent
* Current participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infective endocarditis undergoing open heart surgery with cardio-pulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality (all cause) | 30 days or during index hospitalization
  Overall mortality rate in-hospital, at day 30 or during index hospitalization
Mortality at long-term follow-up | 1 to 5 years
  at 1 to 5 years post-surgery

SECONDARY OUTCOMES:
MACCE | 30 days or during index hospitalization
  Major adverse cardiac and cerebrovascular event rate at day 30 or during index hospitalization.
  Composite of 1.) Cardiac events: (postoperative myocardial infarction, CPR, LCOS/heart failure, repeat cardiac surgery) and/or cerebrovascular events (postoperative stroke, TIA, intracranial hemorrhage)
MACCE at long term follow-up | 1 to 5 years
  Major adverse cardiac and cerebrovascular event rate at 1 to 5 years post-surgery
Sepsis accociated mortatilty | 30 days or during index hospitalization
  Sepsis accociated mortatilty at day 30 or during index hospitalization
Post-operative sepsis | 30 days or during index hospitalization
  Sepsis at day 30 or during index hospitalization
Vasoactive inotropic score | < 72h post-surgery
  The sum of maximum dose rates of inotropes and/or vasopressor medications administered the first 72h post-surgery
Mechanical ventilation time | 30 days or during index hospitalization
  Duration of postoperative invasive/mechanical ventilation post-surgery
Readmission due to IE recurrence | 30 days to 1 year post-surgery
  Recurrence of infective endocarditis after 30 days to 1 year post-surgery
Renal failure | 30 days or during index hospitalization
  Occurence of renal failure (KDIGO criteria)
Dialysis (RRT post-surgery) | 30 days or during index hospitalization
  Occurence of renal failure requiring renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Thielmann, Prof. Dr., Principal Investigator — Department of Thoracic and Cardiovascular Surgery, University Hospital Essen; Jurij Kalisnik, PD. Dr., Principal Investigator — Department of Cardiac Surgery, Hospital Nürnberg, Paracelsus Medical University
Locations (2):
- Germany (2):
  - Department of Cardiac Surgery, Hospital Nürnberg, Paracelsus Medical University, Nuremberg, Bavaria
  - University Hospital Essen, Department of Thoracic and Cardiovascular Surgery, West-German Heart and Vascular Center, University Duisburg-Essen, Essen

REFERENCES:
- [Background] Thornhill MH, Dayer MJ, Nicholl J, Prendergast BD, Lockhart PB, Baddour LM. An alarming rise in incidence of infective endocarditis in England since 2009: why? Lancet. 2020 Apr 25;395(10233):1325-1327. doi: 10.1016/S0140-6736(20)30530-4. No abstract available. PMID 32334690
- [Background] Olmos C, Vilacosta I, Fernandez-Perez C, Bernal JL, Ferrera C, Garcia-Arribas D, Perez-Garcia CN, San Roman JA, Maroto L, Macaya C, Elola FJ. The Evolving Nature of Infective Endocarditis in Spain: A Population-Based Study (2003 to 2014). J Am Coll Cardiol. 2017 Dec 5;70(22):2795-2804. doi: 10.1016/j.jacc.2017.10.005. PMID 29191329
- [Background] Habib G, Erba PA, Iung B, Donal E, Cosyns B, Laroche C, Popescu BA, Prendergast B, Tornos P, Sadeghpour A, Oliver L, Vaskelyte JJ, Sow R, Axler O, Maggioni AP, Lancellotti P; EURO-ENDO Investigators. Clinical presentation, aetiology and outcome of infective endocarditis. Results of the ESC-EORP EURO-ENDO (European infective endocarditis) registry: a prospective cohort study. Eur Heart J. 2019 Oct 14;40(39):3222-3232. doi: 10.1093/eurheartj/ehz620. PMID 31504413
- [Background] Becher PM, Gossling A, Fluschnik N, Schrage B, Seiffert M, Schofer N, Blankenberg S, Kirchhof P, Westermann D, Kalbacher D. Temporal trends in incidence, patient characteristics, microbiology and in-hospital mortality in patients with infective endocarditis: a contemporary analysis of 86,469 cases between 2007 and 2019. Clin Res Cardiol. 2024 Feb;113(2):205-215. doi: 10.1007/s00392-022-02100-4. Epub 2022 Sep 12. PMID 36094574
- [Background] Sy RW, Kritharides L. Health care exposure and age in infective endocarditis: results of a contemporary population-based profile of 1536 patients in Australia. Eur Heart J. 2010 Aug;31(15):1890-7. doi: 10.1093/eurheartj/ehq110. Epub 2010 May 7. PMID 20453066
- [Background] Heiro M, Helenius H, Hurme S, Savunen T, Metsarinne K, Engblom E, Nikoskelainen J, Kotilainen P. Long-term outcome of infective endocarditis: a study on patients surviving over one year after the initial episode treated in a Finnish teaching hospital during 25 years. BMC Infect Dis. 2008 Apr 17;8:49. doi: 10.1186/1471-2334-8-49. PMID 18419812
- [Background] Mylonakis E, Calderwood SB. Infective endocarditis in adults. N Engl J Med. 2001 Nov 1;345(18):1318-30. doi: 10.1056/NEJMra010082. No abstract available. PMID 11794152
- [Background] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Tleyjeh IM, Steckelberg JM, Murad HS, Anavekar NS, Ghomrawi HM, Mirzoyev Z, Moustafa SE, Hoskin TL, Mandrekar JN, Wilson WR, Baddour LM. Temporal trends in infective endocarditis: a population-based study in Olmsted County, Minnesota. JAMA. 2005 Jun 22;293(24):3022-8. doi: 10.1001/jama.293.24.3022. PMID 15972564
- [Background] Bonaros N, Czerny M, Pfausler B, Muller S, Bartel T, Thielmann M, Shehada SE, Folliguet T, Obadia JF, Holfeld J, Lorusso R, Parolari A, Muller L, Grimm M, Ruttmann-Ulmer E. Infective endocarditis and neurologic events: indications and timing for surgical interventions. Eur Heart J Suppl. 2020 Dec 6;22(Suppl M):M19-M25. doi: 10.1093/eurheartj/suaa167. eCollection 2020 Nov. PMID 33664636